CLINICAL TRIAL: NCT03564873
Title: Concomitant Omacetaxine Mepesuccinate and Azacitidine for Patients With Previously Untreated High Grade Myelodysplastic Syndromes
Brief Title: Omacetaxine + Azacitidine in Untreated Patients With High Grade MDS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-2215.cc
Record Dates: First submitted 2018-06-08; First posted 2018-06-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: High Grade Myelodysplastic Syndromes
Keywords: Omacetaxine; Azacitidine; Previously Untreated; Phase I/II; Dose Escalation; Maximum Tolerated Dose
MeSH Terms: interventions — Homoharringtonine; Clinical Trials, Phase I as Topic; Azacitidine; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Up to 18 patients will be enrolled to one of three cohorts to receive various doses of omacetaxine over a 28 day cycle. Azacitidine will be given at the standard dose over a 28 day cycle.
  Interventions: Drug: Omacetaxine; Drug: Azacitidine
- Phase II (Experimental): Up to 33 patients will be enrolled to receive the maximum tolerated dose (determined in phase I) over a 28 day cycle. Azacitidine will be given at the standard dose over a 28 day cycle.
  Interventions: Drug: Omacetaxine; Drug: Azacitidine

INTERVENTIONS:
Drug: Omacetaxine — Phase I is a dose escalation phase. Patients will be enrolled into one of three cohorts to receive omacetaxine subcutaneously (0.5, 0.75, 1.0, or 1.25 mg/m2) twice daily on days 1 to 7.
  Other Names: Phase 1
  Arms: Phase I
Drug: Azacitidine — Azacitidine will be given at the standard dose and schedule, 75 mg/m2 once daily, on days 1 to 7. The patients will then be monitored for 21 more days ( to complete one 28 day cycle) but no more medication will be administered during those 21 days.
  Other Names: Phase 1
  Arms: Phase I
Drug: Omacetaxine — Phase II is a maximum tolerated dose phase. Phase I will determine the maximum tolerated dose (highest amount that can be safely administered). Patients will receive omacetaxine subcutaneously at the maximum tolerated dose (0.5, 0.75, 1.0, or 1.25 mg/m2) twice daily on days 1 to 7.
  Other Names: Phase 2
  Arms: Phase II
Drug: Azacitidine — Azacitidine will be given at the standard dose and schedule, 75 mg/m2 once daily, on days 1 to 7. The patients will then be monitored for 21 more days ( to complete one 28 day cycle) but no more medication will be administered during those 21 days.
  Other Names: Phase 2
  Arms: Phase II

SUMMARY:
This study will treat patients with previously untreated high grade myleodysplastic syndromes (MDS) with both omacetaxine mepesuccinate and azacitidine.

DETAILED DESCRIPTION:
This is an open-label, phase I/II study for previously untreated patients with high grade MDS using omacetaxine and azacitidine with a small expansion cohort for relapsed and refractory MDS patients. Phase I features dose escalation, where patients will be assigned to one of three cohorts to receive different doses of omacetaxine with the standard dose and schedule of azacitidine, over a 28 day cycle. Phase II features the maximum tolerated dose from the Phase 1 study. An additional expansion cohort of 10 MDS patients who have failed to respond to or responded and relapsed after at least one line of therapy containing a hypomethylating agent therapy will also be accrued.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the following criteria within 14 days prior to the first day of therapy (bone marrow biopsy can be performed 28 days prior to the first day of therapy).

1. Subject must have confirmation of high grade MDS (MDS with excess blasts by WHO criteria) or chronic myelomonocytic leukemia with greater than 5% bone marrow blasts
2. Subjects in the newly-diagnosed Phase 2 cohort must have received no prior treatment with a hypomethylating agent for MDS. Subjects in the relapsed/refractory Phase 2 cohort must have received at least 1 prior line of an HMA-containing regimen. "Refractory" is defined as having received at least four cycles of any HMA or HMA-containing regimen with >5-19% bone marrow blasts. "Relapsed" is defined as having >5-19% bone marrow blasts after having achieved a morphologic remission (≤5% bone marrow blasts) after at least one cycle of any HMA or HMA-containing regimen.
3. Subject must be ≥ 18 years of age
4. Subject must have a projected life expectancy of at least 12 weeks
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status of ≤2
6. Subject must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula
7. Subject must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 3.0 × ULN
   * alanine aminotransferase (ALT) ≤ 3.0 × ULN
   * direct bilirubin ≤ 3.0 × ULN
8. Non-sterile male subjects must use contraceptive methods with partner(s) from time of enrollment and continuing up to 90 das after the last dose of study drug. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug.
9. Female subjects must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting omacetaxine; 2) throughout the entire duration of omacetaxine treatment; 3) during dose interruptions; and 4) for at least 90 days after omacetaxine discontinuation.
10. Subject must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the following criteria:

1. Subject is known to be positive for HIV. HIV testing is not required.
2. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load. Hepatitis B or C testing is not required and subjects with serologic evidence of prior vaccination to HBV (i.e., HBs Ag, anti-HBs+ and anti-HBc-) may participate.
3. Subject has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

   * New York Heart Association heart failure > class 2
   * Renal, neurologic, psychiatric, endocrine, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia
4. Subject exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial or fungal). Patients on antibiotics with controlled systemic symptoms will not be excluded.
5. Subject has uncontrolled diabetes
6. Subject has had a recent major hemorrhage or has a bleeding diathesis associated with a high risk of bleeding
7. Pregnant and breastfeeding females.
8. Subject has a history of other malignancies prior to study entry, except for:

   * Adequately treated in situ carcinoma of the breast or cervix uteri
   * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
   * Prostate cancer with no plans for therapy of any kind
   * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recommended Dose | Start of study to end of study, for up to four years
  Determine the recommended dose of omacetaxine based on the maximum tolerated dose.
Overall Response Rate | Study start date to study end date, or death, whichever comes first, up to 4 years.
  Defined by the proportion of patients who achieve any category of complete remission (CR, includes CR and marrow CR) or partial remission (PR) based on the 2006 International Working Group (IWG) criteria for MDS1.

SECONDARY OUTCOMES:
Overall Survival | Study start date to study end date, or death, whichever comes first, up to 4 years.
  Overall Survival will be defined as the time from administration of the initial dose of omacetaxine and azacitidine until death from any cause. This will be measured using Kaplan-Meier survival analysis curves.
Progression Free Survival | Study start date to study end date, or death, whichever comes first, up to 4 years.
  Progression Free Survival will be defined as the amount of time from administration of the initial dose of omacetaxine and azacitidine that a patient lives with the disease but does not get worse. This will be measured using Kaplan-Meier survival analysis curves.
Duration of Response | Study start date to study end date, or death, whichever comes first, up to 4 years.
  Duration of Response will be defined as Time from documentation of tumor response to disease progression.This will be measured using Kaplan-Meier survival analysis curves.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | Start of study to end of study, up to four years
  Safety and tolerability analysis of omacetaxine and azacitidine will be summarized by dose and severity as assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pollyea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universtiy of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Pollyea DA, Stevens BM, Abbott D, Amaya M, Gutman JA, Kent A, McMahon C, Schwartz M, Smith C, Dell-Martin J, Sohalski C, Ellis A, Haag M, Schowinsky J, Pan Z, Patel SB, Ransom M, Gillen A, Jordan CT, Pietras EM. Omacetaxine and azacitidine for untreated patients with myelodysplastic syndromes and excess blasts: a phase I/II clinical trial. EClinicalMedicine. 2025 Oct 10;89:103546. doi: 10.1016/j.eclinm.2025.103546. eCollection 2025 Nov. PMID 41140451

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT03564873/Prot_SAP_ICF_000.pdf